CLINICAL TRIAL: NCT03164850
Title: Laparoscopic Tactile Imaging in Urogynecologic Surgery
Acronym: LTI
Status: Completed | Type: Observational
Sponsor: Advanced Tactile Imaging, Inc. (Industry)
Collaborators: Princeton Urogynecology (Other)
Responsible Party: Sponsor
Other Study IDs: LTI07
Record Dates: First submitted 2017-03-16; First posted 2017-05-24 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2017-05

CONDITIONS: Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Laparoscopic Tactile Imaging — Provides Tactile feedback during laparoscopic surgery

SUMMARY:
During laparoscopic surgery, video camera becomes a surgeon's eyes since the surgeon uses image from the video camera positioned inside the patient's body to perform the procedure. The greatest limitation is the impairment or complete lack of tactile sensation normally used to assist in surgical dissection and decision making. The Investigator proposes to develop a tactile sensing system, Laparoscopic Tactile Imager (LTI), to be used in urogynecological laparoscopic surgery for tactile imaging and tissue characterization (elasticity, structure, boundaries, blood vessel detection) which will be imposed on the video image at area of interest in real time.

DETAILED DESCRIPTION:
For this study, the investigator identified the sacrocolpopexy as the target procedure for the evaluation of LTI. In the cases of sacrocolpopexy, often performed in conjunction with a hysterectomy, one of the most frustrating elements is the lack of tactile feedback at the level of the sacral promontory. The surgeon needs to open up the peritoneum and dissect the underlying tissue to expose the sacral bony structures and ligament without injury to the surrounding bowel, ureter or vascular structures. Sometimes, the sacral promontory is covered with a fat pad which makes it difficult to visualize the promontory and the "safe" space below the aorta and between the iliac arteries/veins is difficult to discern. A difference that is very easy to appreciate with an open procedure where one can easily palpate through the fatty tissues. That step is very critical for the repair and has the greatest potential for catastrophic error without tactile sensation. Because of the reproducibility of the surgical technique and target anatomy for this portion of the procedure, it was thought the sacral promontory dissection to identify and clear the anterior longitudinal ligament would be appropriate surgical procedure to evaluate the use of LTI.

ELIGIBILITY:
Inclusion Criteria:

1. Stage 2 or greater pelvic organ prolapse;
2. Scheduled pelvic floor surgery.

Exclusion Criteria:

1. Active cancer of the colon, rectum wall, cervix, vaginal, uterus or bladder;
2. Ongoing or prior radiation therapy for abdominal or pelvic cancer;
3. Recent (less than four months) pelvic surgery;
4. Surgically absent rectum or bladder;
5. Significant circulatory or cardiac conditions that could cause excessive risk from the examination as determined by attending physician;
6. Severe abdominal or pelvic adhesions preventing access to pertinent anatomy;
7. Known or suspected bleeding disorder.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women scheduled for pelvic floor surgery
Study Population: Adult female subjects volunteers, scheduled for a pelvic floor surgery will be considered to be enrolled in the pilot clinical study. Conditions precluding patients from participation are listed in the study exclusion below ( Eligibility Criteria) criteria. No patients will be excluded on the basis of age or race. Women younger the age 21 will not be included due to the very low probability of pelvic floor diseased condition in the age.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2016-12-09 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
Imaging Performance (resolution in mm) | up to 24 weeks
  The LTI will restore the missing dimension during laparoscopic surgery - the real time 'sense of touch' for tissues and organs of interest. Imaging resolution is a key parameter for the outcome.
Soft tissue elasticity measurement (Pa) | up to 24 weeks
  LTI allows acquisition of stress+strain data to calculate direct tissue elasticity in Pa.

CONTACTS AND LOCATIONS:
Overall Officials: Heather van Raalte, Principal Investigator — Princeton Urogynecology
Locations (1):
- Princeton Urogynecology, Princeton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Scientific Publications of the study results
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 6 months after closing study will be available in Scientific Publications
Access Criteria: Scientific Publications